CLINICAL TRIAL: NCT01973972
Title: Jump Starting Shared Medical Appointments for Diabetes With Weight Management
Brief Title: Jump Start Shared Medical Appointments for Diabetes With Weight Management
Acronym: Jump Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 13-053
Record Dates: First submitted 2013-10-18; First posted 2013-11-01 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
Keywords: Diabetes; Obesity; Complex Care; Primary Care; Chronic Disease
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Chronic Disease | interventions — Shared Medical Appointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight management/shared medical appointment (WM/SMA) (Experimental): Weight management group visits every 2 weeks for 16 weeks using low-carbohydrate diet followed by group visits every 8 weeks (total of 48 weeks) for weight and diabetes management.
  Interventions: Behavioral: Weight management; Behavioral: Shared medical appointments (SMA)
- Shared medical appointments (SMA) (Active Comparator): Diabetes management group visits every 4 weeks for 16 weeks followed by group visits every 8 weeks (total of 48 weeks) for diabetes management.
  Interventions: Behavioral: Shared medical appointments (SMA)

INTERVENTIONS:
Behavioral: Weight management — Weight management group visits using low-carbohydrate diet followed for weight management.
  Arms: Weight management/shared medical appointment (WM/SMA)
Behavioral: Shared medical appointments (SMA) — Diabetes management group visits for diabetes management.

SUMMARY:
The proposed research will test a novel program that combines intensive weight management with shared (group) medical appointments for patients with diabetes. This research is important because diabetes is increasingly prevalent, it requires complex management by the provider and the patient, and weight loss is a critical component of its management. Adding weight management to shared medical appointments could potentially improve blood sugar control while reducing medications and their side effects such as low blood sugar.

DETAILED DESCRIPTION:
Anticipated Impacts on Veteran's Healthcare: Weight management is an important focus of VA as evidenced by its VA/DoD Clinical Practice Guideline and MOVE! program targeting overweight/obesity. VA is also committed to using group visits to increase the efficiency and effectiveness of health care delivery. The investigators aim to test a novel intervention that combines intensive weight and diabetes management using the SMA platform. This research addresses important missions to VA because diabetes is more prevalent in Veterans than in the general population, and because weight management is more challenging and complex in patients with diabetes. Project Background: SMAs involve groups of patients who share a common chronic condition and meet over time to receive education, self-management enhancement, and medication management to improve clinical outcomes. A systematic review by VA found that SMAs modestly improve glycemia in patients with diabetes. Although these SMA programs sometimes included diet and physical activity counseling, weight management was not a primary goal, and weight typically was not reduced. Instead, medication intensification was the primary strategy for improving glycemia, and this strategy can lead to weight gain.

For overweight patients with diabetes, weight loss is first-line therapy because it can improve glycemic control and because excess weight leads to poorer outcomes. Moreover, many antiglycemic medications cause weight gain and hypoglycemic events, which may counteract the potential macrovascular benefits of glycemic control. Dietary interventions, however, can lower weight and improve glycemic control while reducing antiglycemic medication needs and, therefore, subsequent risk for hypoglycemic episodes.

In prior research, the investigators induced weight loss and improved glycemic control while decreasing antiglycemic medications. A combination of an intensive weight management program with the diabetes management offered in SMAs has potential to further improve diabetes outcomes, reduce complications, decrease costs and increase health-related quality of life. Such a combined intervention is ideal for patients with diabetes because of their unique dietary considerations, and their need for careful glycemic and medication management during weight loss. Project Objectives: The investigators will examine whether an intensive, group-based weight management program followed by an SMA intervention (WM/SMA arm) is comparably effective (non-inferior) to the SMA intervention alone for improving glycemic control while using less antiglycemic medication and resulting in fewer hypoglycemic events and lower healthcare costs. Project Methods: 308 overweight VA outpatients with uncontrolled (hemoglobin A1c 8.0% or 7.5% or greater for those under 50) type 2 diabetes will participate in this RCT. Similar to prior SMAs, the SMA visits will occur every 4 weeks for 16 weeks and then every 8 weeks for 32 weeks for a total of 9 visits. Sessions will be led by a physician and trained interventionists, and will include educational topics related to diabetes management (including diet and physical activity), self-management training, and medication adjustment. Similar to the investigators' prior weight management trials, the WM/SMA group will meet every 2 weeks for 16 weeks and then every 8 weeks for 32 weeks for a total of 13 visits. The weight management program will focus on a low carbohydrate dietary pattern because of its potential to lower glycemia, leading to reduced antiglycemic medication needs. After 16 weeks, meeting content will shift to the SMA intervention content but weight management will continue to be addressed at the meetings. The primary outcome is glycemic control assessed by hemoglobin A1c assessed at baseline and at 16, 32, and 48 weeks. Secondary outcomes include hypoglycemic events, changes in the antiglycemic medication regimen as assessed by a summary score, weight and healthcare costs. Diabetes-specific health-related quality of life and medication adherence will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes,
* Hemoglobin A1c >= 8.0% or , >= 7.5 for those less than 50
* BMI >= 27 kg/m2,
* Interest in losing weight,
* Agrees to attend regular visits per study protocol,
* Has access to reliable transportation,
* Has a VAMC provider.

Exclusion Criteria:

* Age >= 75 years old,
* Hemoglobinopathy that interferes with measurement of hemoglobin A1c,
* Certain chronic or unstable diseases that may put the participant at increased risk. These include the following:

  * Kidney disease (serum creatinine >1.5 mg/dL in men, >1.3 mg/dL in women),
  * Type 1 diabetes,
  * Unstable CHD (unstable angina, current/active coronary ischemia workup),
  * Blood pressure 160/100 mm Hg,
  * Fasting triglycerides 600 mg/dL,
  * Fasting serum LDL-C 190 mg/dL,
* Pregnancy, breastfeeding, or lack of birth control if premenopausal,
* Dementia, psychiatric illness, or substance abuse that may interfere with adherence (e.g. illness that is currently unstable or resistant to first-line therapy; substance abuse in the past year),
* Enrollment in another research study that might affect the main outcomes of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Yancy, MD MHS, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crowley MJ, Edelman D, Voils CI, Maciejewski ML, Coffman CJ, Jeffreys AS, Turner MJ, Gaillard LA, Hinton TA, Strawbridge E, Zervakis J, Barton AB, Yancy WS Jr. Jump starting shared medical appointments for diabetes with weight management: Rationale and design of a randomized controlled trial. Contemp Clin Trials. 2017 Jul;58:1-12. doi: 10.1016/j.cct.2017.04.004. Epub 2017 Apr 23. PMID 28445783
- [Result] McVay MA, Yancy WS Jr, Bennett GG, Jung SH, Voils CI. Perceived barriers and facilitators of initiation of behavioral weight loss interventions among adults with obesity: a qualitative study. BMC Public Health. 2018 Jul 11;18(1):854. doi: 10.1186/s12889-018-5795-9. PMID 29996812
- [Result] Yancy WS Jr, Crowley MJ, Dar MS, Coffman CJ, Jeffreys AS, Maciejewski ML, Voils CI, Bradley AB, Edelman D. Comparison of Group Medical Visits Combined With Intensive Weight Management vs Group Medical Visits Alone for Glycemia in Patients With Type 2 Diabetes: A Noninferiority Randomized Clinical Trial. JAMA Intern Med. 2020 Jan 1;180(1):70-79. doi: 10.1001/jamainternmed.2019.4802. PMID 31682682
- [Result] Alexopoulos AS, Yancy WS, Edelman D, Coffman CJ, Jeffreys AS, Maciejewski ML, Voils CI, Sagalla N, Barton Bradley A, Dar M, Mayer SB, Crowley MJ. Clinical associations of an updated medication effect score for measuring diabetes treatment intensity. Chronic Illn. 2021 Dec;17(4):451-462. doi: 10.1177/1742395319884096. Epub 2019 Oct 25. PMID 31653175
- [Result] Sagalla N, Yancy WS Jr, Edelman D, Jeffreys AS, Coffman CJ, Voils CI, Alexopoulos AS, Maciejewski ML, Dar M, Crowley MJ. Factors associated with non-adherence to insulin and non-insulin medications in patients with poorly controlled diabetes. Chronic Illn. 2022 Jun;18(2):398-409. doi: 10.1177/1742395320968627. Epub 2020 Oct 25. PMID 33100020

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA)
Started | 127 | 136
Completed | 109 | 117
Not Completed | 18 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA) | Total
Number analyzed (Participants) | 127 | 136 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.1) | 60.4 (8.3) | 60.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 110 | 125 | 235
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 64 | 79 | 143
  White | 60 | 52 | 112
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 127 | 136 | 263
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 9.0 (1.3) | 9.2 (1.3) | 9.1 (1.3)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 35.6 (5.4) | 35.0 (4.8) | 35.3 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: measure of glycemic control
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA)
Number analyzed (Participants) | 127 | 136
percentage of glycosylated hemoglobin | 8.2 (1.6) | 8.3 (1.4)

2. Secondary Outcome: Hypoglycemic Events
Description: All episodes of hypoglycemia will be recorded by participants on provided standard log forms, noting the date, time, duration, symptoms, treatment received, and concurrent blood glucose. Participants will additionally be asked if they received medical attention for hypoglycemia, and the details if so, since the last assessment. Only one episode will be counted per 24 hours. Serious episodes, defined as <50 mg/dL or 50-69 mg/dL and requiring assistance, will supersede minor episodes in this case.
Time Frame: through 48 weeks
Measure: Mean (95% Confidence Interval); unit: events
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA)
Number analyzed (Participants) | 127 | 136
events | 3.2 [2.1 to 4.4] | 6.6 [4.5 to 8.6]

3. Secondary Outcome: Medication Effect Score
Description: Antiglycemic medications, dosages, and schedules will be assessed carefully with the participant and updated at each visit. A Medication Effect Score (MES), based on the potencies and dosages of the medications in a patient's regimen, was devised to reflect the overall intensity of antiglycemic medication. The MES is calculated as the percentage taken of the maximum dose multiplied by the expected hemoglobin A1c lowering effect for each of a participant's medications, which are then summed. Its range is 0 to infinite, with higher scores meaning higher diabetes medication requirement.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA)
Number analyzed (Participants) | 127 | 136
units on a scale | 2.2 (1.5) | 2.7 (2.0)

4. Secondary Outcome: Weight
Description: weight by electronic scale
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA)
Number analyzed (Participants) | 127 | 136
kg | 104.3 (20.3) | 108.0 (19.5)

5. Secondary Outcome: Estimated Costs of Intervention Strategies
Description: Estimates of intervention costs, utilities, direct and indirect costs using market lab cost estimates
Time Frame: through 48 weeks
Measure: Mean (95% Confidence Interval); unit: U.S. dollars
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA)
Number analyzed (Participants) | 127 | 136
U.S. dollars | 1513.42 [1451.34 to 1575.49] | 1264.49 [1204.39 to 1324.59]

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Weight Management/Shared Medical Appointment (WM/SMA) | Shared Medical Appointments (SMA)
All-Cause Mortality (participants affected / at risk) | 2/127 | 2/136
Serious Adverse Events (participants affected / at risk) | 27/127 | 27/136
Other Adverse Events (participants affected / at risk) | 12/127 | 9/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Management/Shared Medical Appointment (WM/SMA) (N=127) | Shared Medical Appointments (SMA) (N=136)
chest pain/URI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
carotid endarterectomy (Vascular disorders) | 1 (1) | 0 (0)
percutaneous coronary intervention (Cardiac disorders) | 1 (1) | 0 (0)
hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1)
pancreatitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
chest pain/GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemetemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
bedbug infestation (Infections and infestations) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 2 (2) | 0 (0)
angioedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hand injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
pacemaker replacement (Cardiac disorders) | 1 (1) | 0 (0)
gallbladder surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
joint replacement (Surgical and medical procedures) | 2 (2) | 1 (1)
urologic surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
death/cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 2 (2) | 0 (0)
severe hypertension (Vascular disorders) | 1 (1) | 0 (0)
stroke (Vascular disorders) | 2 (2) | 0 (0)
death/esophageal tear (Gastrointestinal disorders) | 1 (1) | 0 (0)
coronary catheterization (Cardiac disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
heart attack (Cardiac disorders) | 0 (0) | 2 (2)
congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
angina (Cardiac disorders) | 0 (0) | 2 (2)
pacemaker firing (Cardiac disorders) | 0 (0) | 1 (1)
death/heart attack (Cardiac disorders) | 0 (0) | 1 (1)
coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 2 (2)
hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
bacterial peritonitis (Infections and infestations) | 0 (0) | 1 (1)
flu-like illness (Infections and infestations) | 0 (0) | 1 (1)
coccyx injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
arm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
urinary obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
prostate cancer (Surgical and medical procedures) | 0 (0) | 1 (1)
lumbar fusion (Surgical and medical procedures) | 0 (0) | 1 (1)
death/stroke (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Management/Shared Medical Appointment (WM/SMA) (N=127) | Shared Medical Appointments (SMA) (N=136)
hypomagnesemia (Endocrine disorders) | 12 (15) | 9 (11)

LIMITATIONS AND CAVEATS:
Original target N not reached due to limited eligible and interested patients. Updated sample size calculation assuming 15% attrition and 1.4% standard deviation for hemoglobin A1c yielded N=254 for 80% power for the non-inferiority hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT01973972/Prot_SAP_000.pdf